CLINICAL TRIAL: NCT01216657
Title: An Open-label, Uncontrolled Phase II Trial of Single Agent Sunitinib (SU 11248) for Patients With Chemo-refractory Metastatic Melanoma
Brief Title: Trial of Single Agent Sunitinib for Patients With Chemo-refractory Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S379 SUMA
Record Dates: First submitted 2010-04-12; First posted 2010-10-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Chemo-refractory Melanoma
Keywords: melanoma; sunitinib
MeSH Terms: conditions — Melanoma | interventions — Sunitinib

ARMS (1):
- sunitinib (Experimental): 50 mg Sunitinib daily for 4 weeks, then 2 weeks without treatment
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50 mg oral, daily, for 4 weeks, then 2 weeks without treatment, repeat at d43

SUMMARY:
Sunitinib is a novel small molecule receptor tyrosine kinase inhibitor with direct antitumor effects as well as antiangiogenetic activity. Preclinical and clinical data for Sunitinib and data about angiogenesis and growth regulation in melanoma suggest the activity of Sunitinib in melanoma. This study will investigate the efficacy, safety and tolerability of Sunitinib as palliative treatment in chemo-refractory metastatic melanoma.

DETAILED DESCRIPTION:
This is a single agent 2-step phase 2 study with a one-year follow-up to evaluate the antitumor activity of Sunitinib administered in treatment cycles of 6 weeks duration (4 weeks treatment and 2 weeks rest) in patients with chemo-refractory melanoma. If the first step shows sufficient efficacy and tolerability the study will continue to step 2. Treatment will continue for 9 months or until disease progression or until intolerable adverse events occur. Subsequently the patients will be followed up for 1 year. Tumor assessment will be performed at baseline, at the end of cycle 1,2,3 and subsequently at the end of every uneven cycle (5,7,9,…).

A total of 40 patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and older.
* Diagnosis of unresectable (Stage III) or metastatic (Stage IV), histologically or cytologically proven, melanoma without clinically meaningful surgical or radiotherapeutical options except for mucosal or ocular origin of the primary tumor.
* Subjects must have completed a first or second line chemotherapy or be progressed under chemotherapeutic treatment. The previous treatment must have included DTIC alone or in combination
* Performance status of 0 to 2 on the ECOG scale
* Life expectancy > 12 weeks.
* Patients must be able to swallow Sunitinib capsules.
* Evidence of measurable disease according to the RECIST criteria
* Prior radiation therapy allowed if completed at least 2 weeks and any major surgery allowed if completed at least 4 weeks prior to first dose of Sunitinib.
* Resolution of all acute toxic side effects of prior therapy or surgical procedures to grade < 1 NCI-CTC (except for laboratory values).
* Adequate organ function including the following:

  * platelets > 100 x 109/L
  * hemoglobin > 8 g/dl
  * absolute neutrophils count (AGC) > 1.5 x 109/L.
* Hepatic:

  * bilirubin <=1.5 times upper limit of normal (ULN)
  * aspartate transaminase (AST) and alanine transaminase (ALT) <=2.5 times normal (AST and ALT <=5.0 times normal is acceptable if liver function abnormalities are due to underlying malignancy).
* INR < 1.5 or a PTT within normal limits.
* Subjects must not have any evidence of a bleeding diathesis.
* Renal:

  * Serum creatinine < 1.5 x ULN
  * serum calcium < 1.2 mg/dl.
* Pancreatic:
* Serum lipase and amylase within normal range.
* Signed and dated informed consent

Exclusion Criteria:

* Prior treatment with ras-raf-MEK-ERK signaling pathway inhibitors (including trastuzumab, sorafenib, farnesyl transferase inhibitors or MEK inhibitors), or treatment with drugs which target VEGF (such as bevacizumab).
* Radiotherapy, except palliative radiotherapy during study participation as described.
* Known active infection (i.e. HIV, chronic hepatitis B or C, at the discretion of the investigator)
* History of organ allograft or stem cell transplantation.
* Coexisting second malignancy (excluding basal or squamous cell carcinoma of the skin, superficial bladder cancer and in situ carcinoma of the cervix with no evidence of recurrence) or history of prior malignancy
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (> hemicolectomie or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis.
* Current history of chronic diarrhea defined as persisting diarrhea for more than 3 weeks at study entry due to any reason.
* Any of the following events prior to starting the trial treatment: *clinically evident congestive heart failure, as defined by New York Health Association (NYHA) > class II

  * Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2
  * Atrial fibrillation of any grade, or prolongation of the QTc interval to >450 msec for males or >470 msec for females.
* Subjects on beta-blockers and digoxin must be monitored closely
* QT-interval > 450 msec
* Risk factors for torsade-de-pointes-tachycardia (i.e.. Hypokalaemia, congenital Long-QT-syndrome)
* Active coronary artery disease or ischemia (myocardial infarction within the last 6 months prior to study entry)
* Coronary/peripheral artery bypass graft
* Cerebrovascular accident or transient ischemic attack
* Active disseminated intravascular coagulation, or history of clinically significant bleeding within the past 6 months, including gross hemoptysis or haematuria, or underlying coagulopathy
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with trial participation or trial drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.
* Participation in any other clinical trial within the last 3 weeks.
* Pregnant or lactating women.
* Known allergic/hypersensitivity reaction to any of the components of the treatment, or known drug abuse/alcohol abuse.
* Active CNS metastatic or meningeal tumors.
* Patients with seizure disorders requiring medication (such as antiepileptics, the use of carbamazepine, phenytion an phenobarbital is prohibited).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
clinical benefit rate cycle 1-3 | tumor assessment every 6 weeks
  clinical benefit rate defined as a CR + PR + SD > 4 months duration
clinical benefit rate cycle 4 and more | tumor assessment every 12 weeks
  clinical benefit rate defined as a CR + PR + SD > 4 months duration

SECONDARY OUTCOMES:
response rate cycle 1-3 | tumor assessment every 6 weeks
  response rate defined as CR+PR
progression free survival | follow-up one year
overall survival | follow-up for one year
response rate cycle 4 and more | every 12 weeks
  response rate defined as CR+PR

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jäger, Prof. Dr., Principal Investigator — Krankenhaus Nordwest
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany